CLINICAL TRIAL: NCT07386990
Title: The Type of Cardioplegia and Cardiometabolic Impact - a Prospective Randomized Trial in Patients Undergoing CABG
Brief Title: Cardioplegic Protection of the Heart
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2021-01728
Record Dates: First submitted 2026-01-28; First posted 2026-02-04 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Bypass Graft (CABG); Cardioplegia; Cardiopulmonary Bypass; Perioperative Myocardial Injury

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Buckberg cardioplegia (Experimental)
  Interventions: Drug: Modified Buckberg cardioplegic solution
- St Thomas´ cardioplegia (Active Comparator)
  Interventions: Drug: Modified St Thomas´ cardioplegic solution

INTERVENTIONS:
Drug: Modified Buckberg cardioplegic solution — Study subjects randomized to this study group will receive Modified Buckberg cardioplegic solution during coronary artery bypass grafting operation.
  Arms: Buckberg cardioplegia
Drug: Modified St Thomas´ cardioplegic solution — Study subjects randomized to this study group will receive Modified St Thomas hospital´s cardioplegic solution during coronary artery bypass grafting operation.
  Arms: St Thomas´ cardioplegia

SUMMARY:
This study seek to compare two different solutions used to protect the heart during cardiac surgery. 40 adult patients planned for coronary artery bypass surgery with cardiopulmonary bypass machine assistance will be included in the study. Blood samples from the first 48 hours after surgery will be analyzed together with physical data, x-ray-results, ecg and general outcome after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for non urgent, single procedure coronary artery bypass grafting surgery at Skåne university hospital in Lund Sweden

Exclusion Criteria: *Heart failure (=Left ventricular ejection fraction less than 40 %).

* Moderate and severe aortic valve insufficiency.
* Type 1 diabetes.
* Renal insufficiency (=estimated glomerular filtration rate <60 mL/min/1,73m2)
* Not communicating in Swedish language.
* Previous cardiac surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2021-11-18 (Actual); Study Completion 2025-04-29 (Actual)

PRIMARY OUTCOMES:
CKMB | 48 hours after surgery (cross clamp release)
  Peak plasma levels of Creatin kinase muscle brain 0,18-300 µg/L

SECONDARY OUTCOMES:
hs-cTnT | 48 hours after surgery (cross clamp release)
  peak level of plasma hig sensitive cardiac Troponin T after surgery 3 - 10 000 ng/L
hs-cTnI | 48 hours after surgery (cross clamp release)
  peak plasma level of high sensitive cardiac Troponin I after surgery 2,50-25 000 ng/L
Pacemaker | two hours after aortic cross clamp release
  Rate of required use of temporary pacemaker after aortic cross clamp release
DC cardioversion | during the surgical procedure in the operating room
  Rate of required use of direct current cardioversion to treat arrythmia after aortic cross clamp release
Cardiometabolic protein profile | 2 hours after surgery
  Levels of 92 cardiometabolic proteins analyzed with proximity extension assay technique before and two hours after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Snejana Hyllén, MD, Assistant Professor, Principal Investigator — Region Skåne
Locations (1):
- Cardiothoracic surgery department, Skåne university hospital, Lund, Lund, Sweden

DOCUMENTS (1):
  • Informed Consent Form (2021-06-01): https://cdn.clinicaltrials.gov/large-docs/90/NCT07386990/ICF_000.pdf